CLINICAL TRIAL: NCT04273243
Title: Long-Term Follow-Up of AT-GTX-501 scAAV9 Gene Transfer in Subjects With CLN6 Batten Disease
Brief Title: Long-Term Follow Up of CLN6 Batten Disease Subjects Following Gene Transfer
Status: Active, not recruiting | Type: Observational
Sponsor: Emily de los Reyes (Other)
Responsible Party: Sponsor-Investigator, Emily de los Reyes, Dr. Emily De Los Reyes, Nationwide Children's Hospital
Organization: Nationwide Children's Hospital (Other)
Other Study IDs: AT-GTX-501-02
Record Dates: First submitted 2020-02-14; First posted 2020-02-18 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: CLN6; Batten Disease
Keywords: Neuronal ceroid lipofuscinosis; NCL; Gene Transfer; vLINCL6
MeSH Terms: conditions — Neuronal Ceroid-Lipofuscinoses

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — During the study, blood samples will be taken for routine lab tests and future tests for safety, effectiveness, or other research assessments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Subjects who received AT-GTX-501 gene transfer: Subjects with CLN6 Batten disease who previously received AT-GTX-501 in the preceding study (Study AT-GTX-501-01).
  Interventions: Genetic: AT-GTX-501

INTERVENTIONS:
Genetic: AT-GTX-501 — No study drug is administered in this study. Subjects who received AT-GTX-501 in a previous trial will be evaluated in this trial for long-term safety and efficacy.

SUMMARY:
This is a long-term safety and efficacy study in subjects with CLN6 Batten disease who previously received a single intrathecal administration of AT-GTX-501.

DETAILED DESCRIPTION:
This is a long-term safety and efficacy study in subjects with CLN6 Batten disease (also know as variant late infantile neuronal ceroid lipofuscinosis associated with mutation(s) in the CLN6 gene [vLINCL6] disease),who previously received a single intrathecal administration of AT-GTX-501. The assessments described in this long-term follow-up (LTFU) study (AT-GTX-501-02) are performed following and in addition to the initial 2 years of post-treatment assessments in the treatment study (AT-GTX-501-01). In this LTFU study, subjects complete safety and efficacy assessments throughout the study's 3-year duration. Combining the duration of the initial treatment study and this LTFU study, the overall duration reflects a follow-up period up-to 5 years since gene transfer via AT-GTX-501.

The primary outcome for this study is to assess the long-term safety of AT-GTX-501 in subjects with CLN6 Batten disease.

The secondary outcome measure of this study is to assess the long-term efficacy of AT-GTX-501 in subjects with CLN6 Batten disease.

ELIGIBILITY:
Inclusion Criteria:

* Subject received AT-GTX-501 (scAAV9.CB.CLN6) in the study "Phase I/IIa Gene Transfer Clinical Trial for Variant Late Infantile Neuronal Ceroid Lipofuscinosis, Delivering the CLN6 Gene by Self-Complementary AAV9."
* Subject completed or prematurely discontinued from the study "Phase I/IIa Gene Transfer Clinical Trial for Variant Late Infantile Neuronal Ceroid Lipofuscinosis, Delivering the CLN6 Gene by Self-Complementary AAV9."
* Subject has a legally authorized representative who has provided written informed consent and authorization for use and disclosure of personal health information or research-related health information.

Exclusion Criteria:

* None

Min Age: 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The subject population in this Long-Term Follow Up study consists of subjects with CLN6 Batten disease who previously received AT-GTX-501 in the preceding study (AT-GTX-501-01).
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2020-01-24 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Long-term safety assessment based on Adverse Events (AEs) | up to 3 years
  All AEs that occur during this study will be classified as treatment-emergent adverse events (TEAEs), as AT-GTX-501 was previously received by all subjects in this study.

SECONDARY OUTCOMES:
Hamburg Scale | up to 3 years
  The Hamburg scale is an established tool to capture the rate of decline or regression. From the Hamburg Scale, the individual motor and language scores and the motor plus language aggregated score will be summarized.

CONTACTS AND LOCATIONS:
Overall Officials: Emily de los Reyes, MD, Principal Investigator — Nationwide Children's Hospital
Locations (1):
- Nationwide Children's Hosptial, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No